CLINICAL TRIAL: NCT04130659
Title: Open, Comparative Study To Evaluate The Performance And Safety Of The Medical Device Marial® In Association With Proton-Pump Inhibitors Versus PPI Alone In Patients Affected By Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Performance and Safety of the MARIAL® in Association With PPI Versus PPI Alone
Acronym: GENYAL®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nekkar Lab Srl (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEK/MD/0119; 2019-004062-17 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Medical Device; Proton-pump inhibitor; Gastroesophageal Reflux Disease; Magnesium Alginate; Mucosal protective agent
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, comparative, multicenter trial with two parallel groups of patients. At the end of the 28-day (± 1) 1st study period, patients will be included in an open-label, non-comparative follow-up (2nd study period) and treated with MARIAL® for additional 5 months from baseline.
Masking Description: Neither the patients nor the Investigator will be blinded to the treatment to which the patients will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MARIAL® and PPI; Follow-up period: MARIAL® alone (Experimental): Period 1, open comparative phase: MARIAL® and PPI administered from day 1 to day 28.
  Period 2, open non comparative follow up: MARIAL® alone administered from day 29 to month 6.
  Interventions: Combination Product: MARIAL® + PPI (generic Omeprazole); Device: MARIAL® alone
- PPI alone; Follow-up period: MARIAL® alone (Active Comparator): Period 1, open comparative phase: PPI alone administered from day 1 to day 28.
  Period 2, open non comparative follow up: MARIAL® alone administered from day 29 to month 6.
  Interventions: Drug: PPI alone (generic omeprazole); Device: MARIAL® alone

INTERVENTIONS:
Combination Product: MARIAL® + PPI (generic Omeprazole) — MARIAL® administration: 1 stick twice daily after meals from day 1 to 28.
  Omeprazole administration: 20 mg cps once daily from day 1 to day 28
  Arms: MARIAL® and PPI; Follow-up period: MARIAL® alone
Drug: PPI alone (generic omeprazole) — Omeprazole administration: 20 mg cps once daily from day 1 to day 28
  Arms: PPI alone; Follow-up period: MARIAL® alone
Device: MARIAL® alone — MARIAL® administration: 1 stick twice daily after meals from day 29 to month 6.

SUMMARY:
Many patients with acid reflux disease do not improve with regular doses of proton pump inhibitors (e.g., omeprazole). The goals of this clinical trial is the to see if taking MARIAL®, in combination with omeprazole, for one month improves symptoms of acid reflux disease compared to taking omeprazole alone.

Furthermore, this study will verify the effectiveness of MARIAL® as a maintenance treatment for the next five months.

This trial is called by the registered name GENYAL®.

DETAILED DESCRIPTION:
This is an open-label, comparative, multicenter study with two parallel groups of patients. The clinical trial has the registered name GENYAL® and will be conducted at five clinical sites.

The study population will include patients affected by gastroesophageal reflux disease (GERD) with a diagnosis of Los Angeles Classification System Grade A reflux esophagitis confirmed by gastroscopy (performed within 1 month prior to baseline) and clinical symptoms in the past 2 weeks.

Patients will be randomized to receive MARIAL® (E-Gastryal®+Magnesium Alginate) plus omeprazole versus omeprazole alone (1 month) followed by Marial® alone for an additional 5 months. The products will be administered following the respective Summary of Product Characteristics. The Investigators chosen the number of rescue medicine used (tablets of Gaviscon®) as a primary efficacy outcome to measure the performance between the two groups. The study will enroll 110 patients.

MARIAL® is a class IIa medical device that is already marketed in several EU countries. It is a combination of E-Gastryal® (hyaluronic acid, hydrolyzed keratin, tara gum, xantan gum, purified water) and magnesium alginate (MgAlg). It has been proven to actively regenerate damaged tissues through its repair and regenerative properties on the mucous membranes and its mucoadhesive and film-forming properties, which prolong the contact time with the mucous membranes and consequently improve their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, both aged ≥ 18 to ≤ 65 years.
* Diagnosis of GERD Grade A esophagitis on Los Angeles Classification System grades reflux esophagitis by:

  * gastroscopy (done within 1-month prior baseline).
  * episodic heartburn and/or acid regurgitation (at least 3 times per week in the last 2 weeks);
* Body mass index of ≥ 18.5 to ≤ 36 kg/m2.
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.
* Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

* Intake of PPI or Marial® during the last 28 days before the start of the study.
* Intake of systemic glucocorticoids or non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2-inhibitors (≥ 3 consecutive days per week) during the last 28 days before the start of the study; except regular intake of enteric coated aspirin dosages up to 150 mg/d.
* Previously underwent acid-lowering surgery or other surgery of the oesophagus and/or upper gastrointestinal tract (excluding appendectomy, cholecystectomy and polypectomy).
* History of co-existing disease that affects the esophagus (e.g. Barrett's esophagus, Zollinger-Ellison syndrome, esophageal stricture).
* History of active gastric or duodenal ulcers within 3 months of the first dose of the study drug or had acute upper gastrointestinal (GI) bleeding within last 6 months.
* Documented presence of severe renal or hepatic insufficiency (i.e. GOT, GPT elevated over double the normal range).
* Known hypersensitivity to omeprazole, and/or Marial® and/or Gaviscon®.
* Concurrent (or within 30 days of study entry) participation in a clinical trial.
* Females who are pregnant, or planning a pregnancy, or lactating. Females of child bearing potential not using reliable methods of birth control.
* Clinically significant laboratory abnormality or disease which, in the opinion of the Investigator, will create a risk for the patient, or interfere with study results (i.e. GOT, GPT elevated over double the normal range).
* Receiving any of the following drugs within 2 weeks before the baseline: theophylline, bismuth salts, warfarin, phenytoin, tacrolimus, diazepam, cyclosporine, disulfiram, barbiturates, antineoplastic agents, erythromycin, clarithromycin, sucralfate, clopidogrel or protease inhibitors. Benzodiazepines could be allowed only in concomitance with the endoscopy.
* Taking concomitant medications that rely on the presence of gastric acid for optimal bioavailability (e.g. ketoconazole, ampicillin esters or iron salts).
* Drug or alcohol abuse within 12 months of Day 0
* Malignancy (also leukemic infiltrates) within 5 years prior to Day 0 (except for treated basal cell/squamous cell carcinoma of the skin).
* Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (except for intermittent anxiety).
* Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study for its safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Total Gaviscon® tablets consumption by patients using alginate as rescue medication | 28 days
  The 28-day visit will assess the outcome by reviewing the patients' diary card. This diary card records their usage of Gaviscon® tablets and calculates the number of unused Gaviscon® tablets they received during baseline. The consumption of Gaviscon® tablets from baseline to the final visit in the Marial® + PPI group will be compared to that of the PPI-only group.

SECONDARY OUTCOMES:
Reflux Symptoms Index (RSI) | 180 days
  RSI is a nine-item self-administered outcome instrument with a maximum total score of 45. The total score can range from zero to 45, with each item being measured using a 6-point rating scale from no problem (0) to severe problem (5). If the score is greater than 13, the RSI will be clinically significant and indicative of reflux disease.
GERD Impact Scale (GIS) | 180 days
  The GERD Impact Scale (GIS) consists of nine questions that cover acid-related symptoms, chest pain, extra-esophageal symptoms, and how the symptoms affect a patient's daily life, including sleep, work, meals, social occasions, and use of over-the-counter medications. The patient will provide their responses using the following four-point Likert scale; 1=none of the time, 2=a little of the time, 3=some of the time, and 4=all of the time for the seven days leading up to the study visit.
GERD Health-Related Quality of Life (GERD-HRQL) | 180 days
  This study employs the 10-item version of the GERD-HRQL questionnaire (Velanovich, V. Diseases of the Esophagus, 2007), which measures intensity and frequency of heartburn, difficulty in swallowing, bloating, and burden of GERD medications. . Responses are rated on a scale of 1 to 5. 0 = No symptoms, 1 = Noticeable but not bothersome, 2 = Noticeable and bothersome but not occurring every day, 3 = Bothersome on a daily basis, 4 = Bothersome and affecting daily activities, 5 = Incapacitating in terms of daily activities. An additional patient-reported global satisfaction score is not added to the total GERD-HRQL score. Hence, the maximum score for this test is 50 and higher scores indicate more severe symptoms and a reduced health-related quality of life.
Investigator Global Assessment of the Performance (IGAP) | 180 days
  Investigator Global Assessment of the Performance (IGAP) will be scored by Investigator as: 1= very good performance, 2 = good performance, 3 = moderate performance and 4 = poor performance. IGAP will be evaluated at day 28 and day 180, only.
Investigator Global Assessment of Safety (IGAS) | 180 days
  Investigator Global Assessment of Safety (IGAS) will be measured using the following 4-point verbal rating scale:1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAP will be evaluated at day 28 and day 180, only.
Serious Adverse Device Effects (SADE), Serious Adverse Events (SAE), Adverse Device Effects (ADE), Adverse Events (AE), and Device Deficiency (DD) | 180 days
  Serious Adverse Device Effects (SADE), Serious Adverse Events (SAE), Adverse Device Effects (ADE), Adverse Events (AE), and Device Deficiency (DD) will be collected and reported by the investigators during the study period. Their incidence will be assessed based on the change from the baseline.
Esophagogastroduodenoscopy (EGD) | 28 days
  Esophagogastroduodenoscopy (EGD) will be evaluated as exploratory outcome. It is a minimally invasive diagnostic procedure that visualizes the upper part of the gastrointestinal tract down to the duodenum. Prior to the procedure, benzodiazepine will be administered for sedation. EGD will be performed at baseline and on day 28 for the 16 patients included in the Italian site only.
GERD recurrence rate | 150 days
  GERD recurrence rate will be evaluated as an exploratory outcome. The rate of GERD recurrence will be assessed by comparing the change from day 28 to day 180.

CONTACTS AND LOCATIONS:
Overall Officials: Doina Rosu, Principal Investigator — Societatea Civilă Medicală Gados
Locations (5):
- UOC Endoscopia Digestiva Chirurgica Policlinico Gemelli - Universita Cattolica, Roma, Italy
- Romania (4):
  - Cabinet Particular Policlinic Algomed, Timișoara, Timiș County
  - Societatea Civilă Medicală Gados, Timișoara
  - Medlife SA, Timișoara
  - Centrul Medical Salvosan Ciobanca, Zalău

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Kung YM, Hsu WH, Wu MC, Wang JW, Liu CJ, Su YC, Kuo CH, Kuo FC, Wu DC, Wang YK. Recent Advances in the Pharmacological Management of Gastroesophageal Reflux Disease. Dig Dis Sci. 2017 Dec;62(12):3298-3316. doi: 10.1007/s10620-017-4830-5. Epub 2017 Nov 6. PMID 29110162
- [Background] Strugala V, Avis J, Jolliffe IG, Johnstone LM, Dettmar PW. The role of an alginate suspension on pepsin and bile acids - key aggressors in the gastric refluxate. Does this have implications for the treatment of gastro-oesophageal reflux disease? J Pharm Pharmacol. 2009 Aug;61(8):1021-8. doi: 10.1211/jpp/61.08.0005. PMID 19703345
- [Background] Aragona SE, Mereghetti G, Bianchetti M, Mangiavillano B, Zurlo T, Lotti J, La Mantia I, Franca K, Lotti T. Regenerative medicine in the treatment of gastro-esophageal reflux disease and laryngo-pharyngeal reflux. From research to cure. J Biol Regul Homeost Agents. 2017 APR-JUN;31(2 Suppl. 2):207-212. PMID 28702984
- [Background] DeVault K, McMahon BP, Celebi A, Costamagna G, Marchese M, Clarke JO, Hejazi RA, McCallum RW, Savarino V, Zentilin P, Savarino E, Thomson M, Souza RF, Donohoe CL, O'Farrell NJ, Reynolds JV. Defining esophageal landmarks, gastroesophageal reflux disease, and Barrett's esophagus. Ann N Y Acad Sci. 2013 Oct;1300:278-295. doi: 10.1111/nyas.12253. PMID 24117649
- [Background] Aragona SE, Mereghetti G, Ciprandi G. Gastric reflux: the therapeutical role of Marial(R). J Biol Regul Homeost Agents. 2018 Jul-Aug;32(4):969-972. PMID 29687692
- [Background] Hillman L, Yadlapati R, Thuluvath AJ, Berendsen MA, Pandolfino JE. A review of medical therapy for proton pump inhibitor nonresponsive gastroesophageal reflux disease. Dis Esophagus. 2017 Sep 1;30(9):1-15. doi: 10.1093/dote/dox055. PMID 28859358
- [Background] Reimer C, Lodrup AB, Smith G, Wilkinson J, Bytzer P. Randomised clinical trial: alginate (Gaviscon Advance) vs. placebo as add-on therapy in reflux patients with inadequate response to a once daily proton pump inhibitor. Aliment Pharmacol Ther. 2016 Apr;43(8):899-909. doi: 10.1111/apt.13567. Epub 2016 Feb 22. PMID 26909885
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Jones R, Coyne K, Wiklund I. The gastro-oesophageal reflux disease impact scale: a patient management tool for primary care. Aliment Pharmacol Ther. 2007 Jun 15;25(12):1451-9. doi: 10.1111/j.1365-2036.2007.03343.x. PMID 17539985
- [Derived] Spada C, Salvi D, Pecere S, Mangiola F, Varca S, Rosu S, Prateek V, Ciobanca PV, Goldis A, Barattini DF, Costamagna G. E-Gastryal(R) + Magnesium Alginate Plus PPI vs. PPI Alone in GERD: Results from the GENYAL(R) Randomized Controlled Trial. J Clin Med. 2025 Jul 7;14(13):4794. doi: 10.3390/jcm14134794. PMID 40649167